CLINICAL TRIAL: NCT01622777
Title: Phase IIa Randomized Double-blind Placebo-controlled Study to Evaluate the Effect of Rosuvastatin in Diabetic Polyneuropathy
Brief Title: The Effect of Rosuvastatin in Diabetic Polyneuropathy: A Phase IIa Randomized Double-blind Placebo-controlled Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alejandra Guillermina Miranda Diaz (Other)
Responsible Party: Sponsor-Investigator, Alejandra Guillermina Miranda Diaz, Investigator of Cardiovascular Research Unit, University of Guadalajara
Organization: University of Guadalajara (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROSU001
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Diabetic Polyneuropathy
Keywords: Rosuvastatin; Diabetic polyneuropathy; Nerve conduction; Oxidative stress; Nerve growth factor
MeSH Terms: conditions — Diabetic Neuropathies; Hereditary Sensory and Autonomic Neuropathies | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Experimental): 20 mg daily of oral rosuvastatin
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — 20 mg daily of oral rosuvastatin for 12 weeks
  Arms: Rosuvastatin
Drug: Placebo — 100 mg of oral placebo with identical appearance, form and size than rosuvastatin, one tablet daily for 12 weeks
  Arms: Placebo

SUMMARY:
To evaluate the impact of oral rosuvastatin in diabetic polyneuropathy, and the role of lipid peroxidation and nerve growth factor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus
* Glycated hemoglobin <12.0%
* Signing of informed consent
* Presence of an abnormality of nerve conduction study
* Symptoms and signs of diabetic polyneuropathy

Exclusion Criteria:

* Pregnancy and lactation
* Foot ulcers
* Treatment with statins
* Antioxidant drug and/or supplements one month previous to enrolment
* Inability to mobilize
* Renal and/or hepatic failure

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Stage of diabetic polyneuropathy | 12 weeks
Severity of diabetic polyneuropathy | 12 weeks
  Severity according nerve conduction studies
Nerve conduction studies | 12 weeks
Neuropathy symptoms and impairment scores | 12 weeks
Lipid peroxidation | 12 weeks
Nerve growth factor | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto G. Cardona-Muñoz, MD, PhD, Study Director — University of Guadalajara; Luis Miguel Roman-Pintos, MD,PhD, Study Chair — University of Guadalajara; Rogelio Troyo-Sanroman, PhD, Study Chair — University of Guadalajara; María del Pilar Alatorre-Carranza, PhD, Study Chair — Hospital Civil de Guadalajara; Alejandra G. Miranda-Diaz, MD, PhD, Study Director — University of Guadalajara; Jaime Hernandez-Ojeda, MD, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Cardiovascular Research Unit. University of Guadalajara., Guadalajara, Jalisco, Mexico